CLINICAL TRIAL: NCT00381173
Title: A Phase 1 Open-Label Study of the Safety and Feasibility of ZYC300 Administration With Cyclophosphamide Pre-Dosing
Brief Title: A Study of ZYC300 Administered With Cyclophosphamide Pre-Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYC3-002
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-07

CONDITIONS: Breast Cancer; Ovarian Cancer; Prostate Cancer; Colon Cancer; Renal Cancer
Keywords: MGI PHARMA; ZYC3-002; ZYC300; plasmid DNA; cyclophosphamide; Cytoxan; advanced breast cancer; advanced ovarian cancer; hormone refractory prostate cancer; advanced colon cancer; advanced renal cancer; advanced stage malignancies; immune therapy; gene therapy; biologic therapy; T-regulatory cells; cancer vaccine; vaccine; Advanced stage malignancies-ovary, breast, colon, prostate
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Kidney Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Cyclophosphamide & ZYC300 (ZYC300 with cyclophosphamide pre-dosing)

INTERVENTIONS:
Drug: Cyclophosphamide & ZYC300 (ZYC300 with cyclophosphamide pre-dosing) — Patients who meet all entry criteria will be administered 600 mg/m^2 cyclophosphamide intravenously 3 days before each dose of ZYC300. ZYC300 will be administered at 400 micrograms DNA/total dose every two weeks for a maximum of six doses (6 cycles).

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety, and tolerability of administering ZYC300 with Cyclophosphamide (Cytoxan).

DETAILED DESCRIPTION:
This is an open-label study of ZYC300 in the treatment of advanced stage malignancy of the kidney in patients who have not had previous immune-based therapies or treatment of advanced stage malignancies (cancerous growths) of the ovary, breast, colon, or hormone-refractory prostate in patients who have failed at least one but no more than two prior regimens of chemotherapy. Patients who meet all entry criteria will be administered 600 mg/m^2 cyclophosphamide intravenously 3 days before each dose of ZYC300. ZYC300 will be administered at 400 micrograms DNA/total dose every two weeks for a maximum of six doses (6 cycles).

ZYC300 is a plasmid DNA formulated within biodegradable microencapsulated particles. This is the first time that ZYC300 and Cyclophosphamide will be given together. Cyclophosphamide is a chemotherapy drug approved by the FDA that has been used for many years in many different kinds of cancer. In this trial the study drug will be used to boost the immune system. Sometimes the immune system cannot fight infected or abnormal cells because of other cells called T reg cells. The T reg cells limit the immune systems attack on infected or abnormal cells. In this study, the hope is that Cyclophosphamide will inhibit the T regs cells so that the ZYC300 can work better to attack the cancer cells.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, patients must meet the following criteria:

1. Patients with:

   Advanced stage malignancies who have failed treatment, including at least one, but no more than two, prior regimens of chemotherapy: Ovary, Breast, Colon, Hormone Refractory Prostate Cancer (HRPC), and renal.
2. Evidence of measurable disease by clinical or radiographic assessment or by tumor biomarker (ovarian and prostate cancer).
3. Age ≥ 18 years old.
4. A baseline Eastern Cooperative Oncology Group Performance Status of 0 or 1.
5. A life expectancy > 6 months.
6. Adequate hematological function established within 14 days prior to receipt of the first dose of cyclophosphamide, defined as:

   1. Absolute lymphocyte count ≥ 1,000/mm^2
   2. WBC ≥ 3,000/mm^2
   3. Platelet count ≥ 75,000/mm^2
   4. Hemoglobin ≥ 9 g/dL
7. Adequate renal function established within 14 days prior to receipt of the first dose of cyclophosphamide, defined as serum creatinine ≤ 1.5 X upper limit of normal.
8. Adequate hepatic function established within 14 days prior to receipt of the first dose of cyclophosphamide, defined as:

   1. Total bilirubin ≤ 1.5 X upper limit of normal, and
   2. SGOT and SGPT ≤ 2.5X upper limit of normal.
9. An MRI of the brain, if clinically indicated, which is negative for parenchymal central nervous system metastases within 28 days prior to receipt of the first dose of cyclophosphamide. If a patient cannot undergo an MRI because of a medical contraindication, a contrast CT of the brain will be acceptable.
10. A negative pregnancy test (blood or urine) within 14 days prior to first dose of cyclophosphamide (where applicable).
11. Agree to use appropriate contraception from study entry until the end-of-observation visit.
12. A signed informed consent form approved by the Institutional Review Board.

Exclusion Criteria:

Patients cannot participate in the study if any of the following apply:

1. Have a history of parenchymal brain metastases.
2. Have received any of the following within 28 days prior to receiving the first dose of cyclophosphamide:

   1. Chemotherapy
   2. Radiation therapy
   3. Immunotherapy
   4. Systemic immunosuppressive drugs
   5. Glucocorticoids (inhalers for asthma are permitted)
   6. Investigational agent or experimental therapy
3. Have received three or more biologic/targeted therapies, such as monoclonal antibodies and tyrosine kinase inhibitors.
4. Have initiated or reinitiated the use of hormonal agents within 28 days prior to receiving the first dose of cyclophosphamide. These drugs are allowed if treatment was initiated greater than 28 days prior to receipt of the first dose of cyclophosphamide.
5. Have a history of bone marrow or stem cell transplantation.
6. Have a history of treatment with fludarabine, 2-chlorodeoxyadenosine, 2-deoxycoformycin or similar compounds.
7. Have a history of treatment with chronic systemic immunosuppressive drugs.
8. Have an immunologic disorder such as immunodeficiency or other chronic auto-immune disease if deemed to be clinically significant.
9. Have an active systemic infection requiring treatment.
10. Are known to be positive for HIV antibody.
11. Pregnant or lactating.
12. Have a history of alcohol abuse, illicit drug use, or psychiatric disorder that would in the Investigator's opinion jeopardize protocol compliance or compromise the patient's ability to give informed consent.
13. Have had prior ex vivo or in vivo DNA therapy (administration of viral vectors or plasmid DNA formulations) or cancer vaccines.
14. Previous exposure to ZYC300 or amolimogene (HPV E6E7 plasmid; formerly known as ZYC101a).

Please note: There may be additional inclusion/exclusion criteria. The study center will determine if patients meet all of the criteria. If patients do not qualify for the trial, study personnel will explain the reasons. If patients do qualify, study personnel will explain the trial in detail using an IRB-approved informed consent, and answer any questions. Patients can then decide if they wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-11; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility, safety and tolerability of administering ZYC300 intramuscularly every other wk for 6 doses (400 micrograms DNA/total dose) to the study pop. pre-dosed with 600 mg/m^2 cyclophosphamide intravenously 3 days prior to study drug. | Within 14 days and 12 weeks post last dose of study drug (and 16 weeks post last dose for response confirmation, if applicable).

SECONDARY OUTCOMES:
Assess the effect of cyclophosphamide on T reg number and function. Assess the generation of CYP1B1-specific immun. as a result of vac. regimen. Assess the effect of vac. regimen on tumor response, if any, in pat. pop. | Within the first 14 days and at each subsequent visit.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverman, MD, Study Chair — Eisai Inc.
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - M. D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Gribben JG, Ryan DP, Boyajian R, Urban RG, Hedley ML, Beach K, Nealon P, Matulonis U, Campos S, Gilligan TD, Richardson PG, Marshall B, Neuberg D, Nadler LM. Unexpected association between induction of immunity to the universal tumor antigen CYP1B1 and response to next therapy. Clin Cancer Res. 2005 Jun 15;11(12):4430-6. doi: 10.1158/1078-0432.CCR-04-2111. PMID 15958627